CLINICAL TRIAL: NCT06756893
Title: The Effect of Sensory Stimulation Thresholds on the Efficacy of Pulsed Radiofrequency Applied to the Dorsal Root Ganglion in Patients with Chronic Lumbar Radicular Pain
Brief Title: The Effect of Sensory Stimulation Threshold on the Efficacy of Pulsed Radiofrequency Applied to the Dorsal Root Ganglion in Patients with Chronic Lumbar Radicular Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Principal Investigator, Ankara University
Other Study IDs: 2024/766
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Dorsal Root Ganglion; Pulsed Radiofrequency; Chronic Pain; Lumbar Radiculopathy; Lumbar Spinal Stenosis
Keywords: dorsal root ganglion; pulsed radiofrequency; lumbar radiculopathy; pain related disability
MeSH Terms: conditions — Chronic Pain; Radiculopathy; Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dorsal Root Ganglion Pulsed Radiofrequency
  Interventions: Procedure: Dorsal Root Ganglion Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Dorsal Root Ganglion Pulsed Radiofrequency — Using C-arm fluoroscopy, a 22G, 10 cm RF needle with a 5 mm active tip will be directed from lateral to medial towards the vertebral foramen. Once the needle reaches the lateral edge of the pedicle shadow, the C-arm will be adjusted to a lateral view to confirm that the needle is located at the craniodorsal portion of the intervertebral foramen. Sensory stimulation will be delivered through the RF generator at 50 Hz, and paresthesia will be sought in the corresponding dermatome at values between 0.4-0.8 mA.
  After achieving paresthesia, motor stimulation at 2 Hz will be applied, and the location near the DRG will be confirmed if motor stimulation is not elicited at values less than 1.5 times the sensory threshold. Pulsed RF will then be applied for 4 minutes at a setting of 45 V, 20 ms pulse width, and 2 Hz frequency. Following the application, needle will be directed slightly anterior and after appropriate contrast flow, dexamethasone will be injected.

SUMMARY:
Lomber dorsal root ganglion pRF is an interventional treatment options in the treatment of lumbar radicular pain. The goal of this study is to investigate the effect of sensory threshold outcomes on pain severity during dorsal root ganglion pulsed radiofrequency (DRG-pRF). It will also learn effects about disability due to chronic LRP. The main questions it aims to answer are:

Does lower sensory threshold result in lower pain scores and chronic LRP related disability?

Participants will:

Take DRG-pRF procedure for 4 minutes. Visit the clinic at 1. and 3. month for questionnaries.

DETAILED DESCRIPTION:
Lumbar radicular pain is characterized by sharp, stabbing, or throbbing pain radiating to one or more dermatomes. It is a common and challenging condition for clinicians to manage in pain practice. Conservative treatments such as physical therapy, non-steroidal anti-inflammatory drugs, rest, and exercise may fail, leading to chronic pain. In such cases, minimally invasive methods such as epidural steroid injection (ESI) or pulsed radiofrequency (pRF) of the dorsal root ganglion (DRG) may be preferred.

Unlike conventional radiofrequency, pRF does not cause ablation. Due to the intermittent delivery of energy generated by the electric current, the target tissue temperature does not exceed 42°C. This creates a magnetic field that modulates pain without causing neuronal damage.

The DRG, highly sensitive to mechanical compression, is a critical target in radicular pain. There is evidence supporting the efficacy of DRG pRF in chronic lumbar radicular pain. Studies comparing pRF alone or in combination with ESI versus ESI alone have found it effective in providing long-term pain relief. However, despite the increasing body of evidence, studies are lacking on the impact of the proximity of pRF to the target neuronal tissue on clinical outcomes.

The primary aim of this study is to investigate the relationship between the sensory stimulation threshold, indicating the proximity to the target tissue during DRG pRF, and the reduction in Numeric Rating Scale (NRS) scores at the 3-month follow-up. Secondary objectives include examining the relationship between Oswestry Disability Index (ODI) and NRS scores at various assessment time points.

The DRG, highly sensitive to mechanical compression, is a critical target in radicular pain (5,6). There is evidence supporting the efficacy of DRG pRF in chronic lumbar radicular pain. Studies comparing pRF alone or in combination with ESI versus ESI alone have found it effective in providing long-term pain relief (7). However, despite the increasing body of evidence, studies are lacking on the impact of the proximity of pRF to the target neuronal tissue on clinical outcomes.

The primary aim of this study is to investigate the relationship between the sensory stimulation threshold, indicating the proximity to the target tissue during DRG pRF, and the reduction in Numeric Rating Scale (NRS) scores at the 3-month follow-up. Secondary objectives include examining the relationship between Oswestry Disability Index (ODI) and NRS scores at various assessment time points.

ELIGIBILITY:
Inclusion Criteria:

Pain lasting ≥3 months NRS score ≥4 Unilateral pain Diagnosis of spinal stenosis or lumbar disc herniation causing root compression, confirmed by magnetic resonance imaging (MRI) according to appropriate diagnostic criteria and classification Failure of conservative treatment

Exclusion Criteria:

Unwillingness to participate in the study Epidural steroid injection within the past month Uncontrolled psychiatric disorders despite medical treatment Systemic or localized infection signs at the procedure site Severe spinal stenosis Allergy to steroids or contrast agents History of cancer Coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates who visited algology clinic of Ankara University Medicine Faculty Hospitals to DRG-pRF prodecure for chronic LRP.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Postprocedure pain severity at 3th month | From procedure to 3 months after prodecure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at 3 months after interventions. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.

SECONDARY OUTCOMES:
Postprocedure pain severity at 30. min | From procedure to 30 minustes after procedure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at 30. min after interventions at bedside. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.
Postprocedure first month pain severity | From procedure to 1 month after procedure
  Severity of pain will be assessed with Numeric Rating Scale (NRS-11) at 1 month after interventions. NRS-11 is a 11 point likert type scale. Higher scores represent more severe pain.
Postprocedure first month OSWESTRY scores | From procedure to 1 month after procedure
  Disability will be assessed with OSWESTRY Diasability Index at 1 month. OSWESTRY measures pain related lumbar disability. It has 0 minimum and 100 maximum value. Lower scores represent better outcomes.
Postprocedure 3th month OSWESTRY scores | From procedure to 3 month after procedure
  Disability will be assessed with OSWESTRY Diasability Index at 3 month. OSWESTRY measures pain related lumbar disability. It has 0 minimum and 100 maximum value. Lower scores represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Güngör Enver Özgencil, MD, Study Director — Ankara University Medicine Faculty Anesthesiology and Reanimation Department

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared except personal data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 5 years after January 2026
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Cohen SP, Strassels SA, Kurihara C, Lesnick IK, Hanling SR, Griffith SR, Buckenmaier CC 3rd, Nguyen C. Does sensory stimulation threshold affect lumbar facet radiofrequency denervation outcomes? A prospective clinical correlational study. Anesth Analg. 2011 Nov;113(5):1233-41. doi: 10.1213/ANE.0b013e31822dd379. Epub 2011 Sep 14. PMID 21918166
- [Background] Park S, Park JH, Jang JN, Choi SI, Song Y, Kim YU, Park S. Pulsed radiofrequency of lumbar dorsal root ganglion for lumbar radicular pain: A systematic review and meta-analysis. Pain Pract. 2024 Jun;24(5):772-785. doi: 10.1111/papr.13351. Epub 2024 Jan 31. PMID 38294072